CLINICAL TRIAL: NCT06674408
Title: Effects of Proprioceptive and Hand Function Exercises in Management of Acute Adhesive Capsulitis
Brief Title: Proprioceptive Exercises in Acute Adhesive Capsulitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RCRAHS-ISB/REC/MS-PT/01871
Record Dates: First submitted 2024-11-03; First posted 2024-11-05 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Adhesive Capsulitis
Keywords: adhesive capsulitis; frozen shoulder
MeSH Terms: conditions — Bursitis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prioprioceptive exercises (Experimental): Hot packs, mobilization, stretching and strengthening, closed and open chain kinetic exercises, hand function exercises, hand eye coordination exercises
  Interventions: Other: Prioprioceptive group
- Conventional (Active Comparator): Hot packs, mobilization, stretching and strengthening, finger ladder exercise, Codman's pendulum exercise, towel stretch exercise and wand exercises
  Interventions: Other: Traditional physical therapy

INTERVENTIONS:
Other: Traditional physical therapy — Control group included Hot pack over shoulder region for 15 mins. Shoulder AP, PA and inferior glides (Maitland) Grade II, III, IV 30 reps x 3 sets per session, Stretching of levator scapula, upper trapezius, pectoralis major and minor with 15 second hold x 3 reps per session, Strengthening of rotator cuff muscles by manual resistance with 10 second hold x 5 reps x 2 sets per muscle per session, Finger Ladder Exercise, Codman's Pendulum Exercise, Towel Stretch Exercise and Wand Exercises 10 reps x 2 sets per session,
  Patients were assessed for baseline measurements against outcome measures. Patients were given a total of 10 sessions such that 5 sessions per week for the duration of 02 weeks. All patients were reassessed at the end of the 1st and 2nd week of treatment for outcome measures.
  Arms: Conventional
Other: Prioprioceptive group — Experimental group included Hot pack over shoulder region for 15 mins. Shoulder AP, PA and inferior glides (Maitland) Grade II, III, IV 30 reps x 3 sets per session, Stretching of levator scapula, upper trapezius, pectoralis major and minor with 15 second hold x 3 reps per session, Strengthening of rotator cuff muscles by manual resistance with 10 second hold x 5 reps x 2 sets per muscle per session, Plyometric CKC shoulder exercise 10 seconds each x 5 reps x 2 sets per session, CKC exercise on the ball 10 seconds each x 5 reps x 2 sets per session, Open KC exercises 10 seconds each x 5 reps x 2 sets per session, Hand-eye coordination exercises for 30 minutes/per day for 5x/per week, Hand Function Exercises for 30 minutes/per day for 5x/per week.
  Patients were assessed for baseline measurements against outcome measures. Patients were given a total of 10 sessions such that 5 sessions per week for the duration of 02 weeks. All patients were reassessed at the end of the 1st and 2nd week
  Arms: Prioprioceptive exercises

SUMMARY:
The purpose of the study is to explore the effect of proprioceptive and hand function exercises in management of acute adhesive capsulitis. A randomized control trial was conducted at RIH Sihala, DSK Bahria town phase 7 and MRC MIHS Rawalpindi. The sample size was 44 calculated through G-power 3.1. The participants were divided into two interventional groups each having 22 participants. The study duration was six months. Sampling technique applied was convenience sampling for recruitment and group randomization using flip coin method. Only 35 to 50 years participants with acute adhesive capsulitis were included in the study. Tools used in this study are Goniometer, NPRS, SPADI and DASH. Data was collected at baseline, at the end of 1st week and 2nd week. Data analyzed through SPSS version 26.

DETAILED DESCRIPTION:
Adhesive capsulitis is one of the commonly encountered musculoskeletal disorders in physical therapy, and has debilitating effects on quality of life. Adhesive capsulitis has been traditionally classified into freezing, frozen and thawing stages, based on the disease course and natural history. The freezing stage, also known as the acute stage, is characterized by insidious and gradual loss of range of motion along with pain, especially at night. The acute stage lasts from the onset till anywhere from 2 to 9 months depending upon the intervention.

According to a recent systematic review, exercise therapy is beneficial for improving function and range of motion in patients with adhesive capsulitis, although to an uncertain degree of evidence. Another systematic review on occupational therapy interventions in musculoskeletal disorders found strong evidence for range of motion exercises and joint mobilizations when combined with steroid injections.

Hand function assessment is done mainly in neurological conditions and largely ignored in most musculoskeletal disorders of the shoulder and elbow, unless there is direct and significant impairment of the Hand function. However, literature supports the need of proximal stability in order to achieve distal mobility regardless of the activity being gross or fine motor. The physiological basis behind this are supported by electromyography studies showing the facilitation-inhibition effects of motor cortex neurons on spinal motor neuron pools of shoulder and distal upper limb musculature.

Descending commands directly influencing motor output have Corticomotoneuronal cells of the primary motor cortex as one of the sources, connecting monosynaptically with the motor neurons. Corticomotoneuronal cells give divergent outputs to muscles of the distal forelimb muscles, which raises the possibility that a single Corticomotoneuronal cells may represent even more complex output patterns. In addition to the musculature of the wrist and hand, those of the shoulder, elbow and trunk might be included in these complex patterns. For instance, during a reach and prehension task, Corticomotoneuronal cells influence muscles at multiple joints of the forelimb, through co-activation of proximal and distal muscles in coordinated, functional synergies which are in line with performance of different phases of the task.

Furthermore, the kinetic link model advocates for the proximal-to-distal sequencing when attempting to restore function, as efficient motion and muscle activation occur with rehabilitation of the entire neuromuscular system through multi-segment integration, rather than isolated treatment of the primarily involved area. According to the kinetic chain rehabilitation, by performing multi-segment exercises the involved muscles can be activated when facilitated by adjacent segments, developing appropriate shoulder function and motion (irradiation). Decreasing the role of the facilitating segments later in the progression increases the load and functional demand on the shoulder. Kinetic chain shoulder exercises, by employing the natural motor programs of motor control, focus on the neuromuscular system rather than on isolated movement and muscle activation.

Hand function exercises are not a routine part of rehabilitation protocol for management of adhesive capsulitis and literature is scarce for high quality evidence regarding efficacy and uniform dosage of Hand function and proprioceptive exercises to be included in the plan of care. A randomized study found no differences at 12 weeks for outcomes when showing effectiveness of proprioceptive exercises for sub-acromial impingement syndrome. A recent study found significant improvement for functional activity on DASH scale and pain on SPADI in proprioception group compared to conventional treatment for adhesive capsulitis, however no differences were found for range of motion and disability on SPADI in post-treatment analysis. Another study reported greater functional improvements in Maitland and Hand function exercises group, compared to Maitland group alone. However, both groups had home exercises, so the effect is unclear as evidence supports improvements for supervised exercises rather than those done at home.

In both the mentioned studies, no long-term follow up was made and patients were only treated for a period of one month. Furthermore, it is unclear what role other interventions included in the management program played in achieving the outcomes as there is no standard protocol set for adhesive capsulitis. The studies also lacked details on what type of mobilization technique to use alongside, as well as the grades of mobilizations to use. One of the studies had no blinding for treatment group allocation, while the other lacked randomization and did not calculate sample size. Both studies included patients of adhesive capsulitis in the sub-acute stage, therefore the evidence is deficient whether patients in the acute stage will benefit from proprioceptive and Hand function exercises.

Therefore, the current study aims to further explore the effect of proprioceptive and Hand function exercises in management of acute adhesive capsulitis. Incorporating these exercise interventions in the acute stage of adhesive capsulitis may result in timely resolution of the symptoms and lower the risk of progressing to later stages and developing disability. The findings of this study will help in further clearing the effectiveness so that the exercises can be made part of the routine management plan for acute adhesive capsulitis.

ELIGIBILITY:
Inclusion Criteria:

* Painful and limited active and passive glenohumeral ROM
* Freezing or acute stage of adhesive capsulitis
* Positive Coracoid pain and DTPER tests
* Primary adhesive capsulitis/secondary due to diabetes mellitus
* Consenting to participate in the study

Exclusion Criteria:

* Bilateral adhesive capsulitis
* Sub-acute and chronic stages of adhesive capsulitis
* Unstable fractures or surgical fixation in the affected limb
* Rheumatoid arthritis
* Severe joint pain unrelieved by rest
* Osteoporosis
* Radiating pain due to cervical conditions
* Manipulations under anesthesia
* Shoulder conditions such as subacromial pain syndrome, rotator cuff tendinopathy, shoulder bursitis etc.
* Neurological damage due to stroke or Parkinsonism
* Cognitive deficits and not giving consent.

Ages: 35 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2024-05-03 (Actual); Primary Completion 2024-12-03 (Actual); Study Completion 2024-12-03 (Actual)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale | 2nd Week
  Changes from Baseline pain values were taken with the help of Numeric Pain Rating Scale measures level of pain. Scoring is done by selecting a point from zero to ten as the current level of pain. Zero means minimum pain and 10 denotes maximum pain.
Range of motion | 2nd Week
  Changes from Baseline shoulder range of motion taken with the help of universal goniometer

SECONDARY OUTCOMES:
Shoulder Pain and Disability Index | 2nd Week
  Changes from the Baseline shoulder pain and disability was taken with help of Shoulder Pain and Disability Index. Scoring is done by separately scoring pain and disability components and adding the two and then dividing by two. Lower scores mean low disability while higher scores show greater disability.
Disability of Arm, Shoulder and Hand | 2nd Week
  Changes from the Baseline problems with arm, shoulder and hand were taken with the help of Disability of Arm, Shoulder and Hand. Scoring is done by totaling responses and dividing by total number of responses and then subtracting from one and multiplying by twenty-five. Lower scores mean less disability and greater scores mean higher disability.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Affan Iqbal, PhD, Principal Investigator — Riphah International University, Islamabad
Locations (3):
- Pakistan (3):
  - Riphah International Hospital, Islamabad
  - DSK Physio and Rehab, Rawalpindi
  - Margalla Rehab Center, Rawalpindi

IPD SHARING:
Plan to Share IPD: No